CLINICAL TRIAL: NCT01149603
Title: The Destination Therapy Evaluation for Failing Fontan Study (DEFINe Study)
Brief Title: The Destination Therapy Evaluation for Failing Fontan Study
Acronym: DEFINe
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollement
Sponsor: Timothy Icenogle, MD (Other)
Responsible Party: Sponsor-Investigator, Timothy Icenogle, MD, Director of Heart Transplant & VAD, Providence Health & Services
Organization: Providence Health & Services (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G090176
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Failing Fontan Physiology; Failing Fontan; Single-ventricle; Single-ventricle Fontan; Single-ventricle Physiology
Keywords: failing Fontan; single-ventricle; destination therapy; HeartMate II; HMII; cardiac congenital anomaly; ventricular assist device; VAD
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation of the HeartMate II VAD (Experimental): Consenting patients who meet the study inclusion and exclusion criteria will be implanted with a HeartMate II ventricular assist device.
  Interventions: Device: HeartMate II Ventricular Assist Device

INTERVENTIONS:
Device: HeartMate II Ventricular Assist Device — The HeartMate II Left Ventricular Assist Device has been approved by the FDA for use in bridge-to-transplant therapy and destination therapy for patients with endstage heart failure.
  Other Names: HMII, HMII LVAD

SUMMARY:
Purpose: The purpose of the Destination Therapy Evaluation for Failing Fontan Study (DEFINe Study) is to perform a single center physician-investigator led feasibility study to initiate examination of the safety and efficacy of implanting continuous flow circulatory support devices in 20 patients with failing Fontan physiology, not amenable to other surgical or medical therapy and who are not candidates for heart transplantation. Based upon the results of the DEFINe study, consideration would be given to a larger multicenter study. The primary endpoint is survival without a disabling stroke at two years. Safety, functional status, total days alive following hospital discharge and quality of life assessments will be evaluated as secondary endpoints.

Background: Patients born with the congenital anomaly of a single ventricle often undergo Fontan procedures to improve oxygenation and circulation. As the patient matures, the benefits of the Fontan procedures become exhausted. These patients present as young adults with heart failure, and should be considered for heart transplantation. "Failed Fontan" physiology patients are now more commonly surviving into their 30s and 40s due to the advancement in surgical Fontan procedures over the last several decades. Yet, many patients are not appropriate transplant candidates due to progression of pulmonary failure that surpasses the pulmonary vascular resistance limits, end organ failure effects to the liver, and cardiac failure that does not present with left ventricular ejection fractions of less than 25%. Congenital heart disease is considered a higher risk indication for transplantation. Such patients present a complex anatomy, scar tissue from prior procedures, unique pathological states and limited ability to assess hemodynamics.

Methods: Patients with failing Fontan physiology will be evaluated for surgical intervention, heart transplantation or participation in the study for long-term support, known as Destination Therapy (DT). Patients who do not meet the study criteria will be asked to participate in a sub-study to collect patient information. Consenting patients who meet the study criteria will be implanted with a HeartMate II Ventricular Assist Device (VAD) to improve cardiac output. Following VAD implantation, the patient will recover in the hospital, and then discharge to home or an approved facility. Study data will be collected as long as the patient receives VAD support. Placement of the VAD and continuing patient care should improve cardiac output and quality of life for this population of patients born with the congenital anomaly of a single ventricle.

Outcomes: The primary endpoint of the study is to examine survival without a disabling stroke at two years (defined as a score of four or greater on the Modified Rankin Scale). Safety, functional status, total-days-alive following hospital discharge, and quality of life assessments will be evaluated as secondary endpoints.

DETAILED DESCRIPTION:
Study Design:

This is a single center nonrandomized observational study led by the PI. However, patients will be recruited from other centers to participate in this trial. The recruited patients will be ineligible for cardiac transplantation at the referring institution. The study institution will also evaluate the patient for cardiac transplantation. If the patient is determined to be ineligible for transplantation at the study institution, the patient will have met the study inclusion criteria pertaining to two institutional turn downs for transplant. The protocol has been designed this way to attract the proposed 20 study patients, and to allow for a second opinion as to whether the patient is a transplant candidate. The patient may pursue cardiac transplantation at an institution that deems him/her transplant eligible, if applicable.

Those patients who are not candidates for transplantation could then be considered for the proposed research study. Patients will need to sign an informed consent to be screened for the study.

Patients who meet the inclusion and exclusion criteria will be implanted with the HeartMate II VAD and data will be collected as described below in the section "data collection". Patients who fail to meet the study inclusion and exclusion criteria will be asked to participate in a sub-study. The sub-study will collect screening and baseline data, as clinically indicated.

Primary Endpoint:

The primary endpoint is to examine survival without a disabling stroke at two years (defined as a score of four or greater on the Modified Rankin Scale). Patients that reach the primary endpoint of survival without a disabling stroke at two years will be considered a success in this study. The percent of patients that have a successful outcome should be targeted at 80% of patients that survive to 2 years without a disabling stroke in the general Destination Therapy patient population at Providence Sacred Heart Medical Center. The current survival rate is 53% survival at 2 years. Therefore, a primary endpoint of 40% survival (8 out of 20 patients) to 2 years without a disabling stroke is purposed. Data related to freedom from a disabling stroke is roughly based on the work published by Tsukui et al. that showed 33-75% freedom from cerebrovascular accidents at 6 months in differing device groups of patients waiting as bridge-to-transplant candidates.

Secondary Endpoints:

Safety, functional status, total-days-alive following hospital discharge, and quality of life assessments will be evaluated as secondary endpoints. Secondary endpoints will be evaluated throughout the study and at one- and two- year follow-up time points after the last patient has been enrolled into the study. The study is designed to improve quality of life, in addition to length of life.

* Safety will be evaluated for all cause mortality, incidence of serious adverse events, as per the Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) definitions (except for modified bleeding and neurocognitive event definitions), and Incidence of device replacement or device repair due to failure.
* Functional status and hospitalizations will be evaluated by the cardio-pulmonary stress test (V.O2 peak), New York Heart Association class, 6-minute walk test, and total number of days alive out-of-hospital.
* Quality of life will be assessed through the Minnesota Living with Heart Failure and Euro-QOL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age greater than or equal to 18 years
* Appropriate surgical candidate for the HeartMate II LVAD
* Willing to consider treatment with the HeartMate II LVAD
* BSA greater than or equal to 1.2
* Female patients must be using adequate contraceptive methods or be unable to become pregnant (2 years post-menopausal or surgically sterilized)
* Patient has Stage D heart failure for, at least, 60 days despite optimal medical management for at least the last 60 days
* Functional limitation due to heart failure as defined by at least ONE of the following:

  1. A history of a progressive downhill course manifested by a restricted quality of life, or increasing hospital admissions, or increasing medication requirements
  2. Presence of protein losing enteropathy
* Ineligible for cardiac transplantation at Sacred Heart Medical Center and at least one other UNOS approved heart transplant center, in the judgment of that center's multidisciplinary transplant team
* Ability to read, understand and implement the instructions for use for the HeartMate II LVAD

Exclusion Criteria:

* Technical obstacles that pose an inordinately high surgical risk, in the judgment of the investigator
* Uncorrectable acquired coagulopathy
* Primary coagulopathy or platelet disorder, including thrombocytopenia with absolute platelet count < 80k or active state of disseminated intravascular coagulation
* Contraindication to the administration of heparin, warfarin or anti-platelet agents
* Severe intrinsic pulmonary disease in the judgment of the investigator
* On mechanical ventilatory support and unable to be weaned
* Patient is under consideration for reparative cardiac surgery (likely to result in clinical resolution of the heart failure in the judgment of the investigator)
* Prior implantation of an assist device
* Mechanical prosthetic aortic or mitral valve that will not be converted to a bio-prosthesis at time of VAD implantation
* Moderate or severe (>1+) aortic insufficiency as determined by echocardiogram that is not amenable to surgical repair or replacement
* Evidence of severe intrinsic hepatic disease as defined as biopsy proven liver cirrhosis with a likelihood of less than two years survival; or liver enzyme values (AST, ALT or total bilirubin) that are > 3 times the upper limit of normal within 30 days prior to surgery, except if the result of acute heart failure decompensation as determined by the investigator
* Creatinine of > 3.5mg/dl or any form of dialysis within 24 hours prior to surgery
* Stroke within 90 days prior to surgery, or history of cerebral vascular disease with significant (> 80%) extra cranial or intra cranial stenosis documented by carotid doppler study or angiography, without evidence of collateral flow documented by transcranial doppler study
* Alzheimer's disease and/or impaired cognitive function, or any other form of irreversible dementia (or both) that is confirmed by a neurological exam
* Patient has evidence of an untreated abdominal aortic aneurysm ≥ 5 cm as measured by abdominal ultrasound
* Suspected or active systemic infection within 48 hours prior to surgery
* Significant peripheral vascular disease as defined by rest pain or ulceration
* Patient in whom abdominal surgery is planned
* Positive serum pregnancy test, for women of childbearing potential
* Recent history of psychiatric disease or psycho-social maladaptive behaviors (including drug or alcohol abuse) that are likely to impair compliance with the study protocol, in the judgment of the investigator
* Therapy with an investigational intervention at the time of screening, or plan to enroll patient in additional investigational intervention study during participation in this trial
* Patient has a condition, other than heart failure, which would limit survival to less than 2 years
* Patient is eligible for cardiac transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2017-09-19 (Estimated); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Survival to 2 years without a disabling stroke | 2 years
  The primary endpoint is to examine survival without a disabling stroke at two years (defined as a score of four or greater on the Modified Rankin Scale). The percent of patients that have a successful outcome should be targeted at 80% of patients that survive to 2 years without a disabling stroke in the general Destination Therapy patient population at Providence Sacred Heart Medical Center. The current survival rate is 53% survival at 2 years. Therefore, a primary endpoint of 40% survival (8 out of 20 patients) to 2 years without a disabling stroke is purposed.

SECONDARY OUTCOMES:
Safety | 2 years
  Safety will be evaluated for all cause mortality, incidence of serious adverse events, as per the Interagency Registry for Mechanically Assisted Circulatory Support definitions, and incidence of device replacement or device repair due to failure.
Functional Status | 2 years
  Functional status and hospitalizations will be evaluated by the cardio-pulmonary stress test, New York Heart Association class, 6-minute walk test, and total number of days alive out-of-hospital.
Quality of Life | 2 years
  Quality of life will be assessed through the Minnesota Living with Heart Failure and Euro-QOL questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Icenogle, M.D., Principal Investigator — Providence Sacred Heart Medical Center
Locations (1):
- Providence Sacred Heart Medical Center, Spokane, Washington, United States